CLINICAL TRIAL: NCT02624076
Title: A Randomized Controlled Trial of Acupuncture Versus Expectant Management in Women With Unexplained Infertility
Brief Title: Acupuncture for Unexplained Subfertiliy
Acronym: AURIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiaoke Wu, Director of obstetrics and gynecology, First Affiliated Hospital of Heilongjiang Chinese Medicine University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AURIS2015
Record Dates: First submitted 2015-11-24; First posted 2015-12-08 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Unexplained Infertility
Keywords: unexplained infertility; Acupuncture
MeSH Terms: interventions — Acupuncture Therapy; Watchful Waiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture plus expectant management (Experimental)
  Interventions: Other: Acupuncture; Other: expectant management
- expectant management (Active Comparator)
  Interventions: Other: expectant management

INTERVENTIONS:
Other: Acupuncture — semi-fixed protocol will be used including four local core points; conception vessel (CV) 3, CV 6, and stomach (ST) 29 bilaterally and four in the leg/feet; spleen (SP) 6, and SP 9 bilaterally. The core points CV 3, CV 6, ST 29, SP 6, and SP 9 are thereafter connected to electrical stimulator (Hwoto, China) and stimulated with low-frequency, 2Hz, 0.5 ms
  Arms: Acupuncture plus expectant management
Other: expectant management — one initial counselling session, an information leaflet on timed intercourse, access to a telephone helpline for queries and ad hoc support on demand from the fertility clinic over a period of 4 months post randomization.

SUMMARY:
Infertility affects one in six couples. In a quarter of them, routine tests of semen quality, ovulation or tubal patency fail to reveal any abnormalities and the cause of infertility is unexplained. Acupuncture is being increasingly used by couples with all types of infertility and initial trials have suggested that it could be potentially beneficial in some cases. A number of systematic reviews of acupuncture in IVF have shown conflicting results, but there is no evidence to inform best practice in unexplained infertility. In addition, as an intervention, acupuncture is not cost neutral as it involves multiple visits for treatment sessions delivered by a skilled practitioner. Thus, while acupuncture could have the potential to increase live birth rates in women with unexplained infertility, the clinical and cost effectiveness of acupuncture needs to be confirmed in the context of a large randomized controlled trial.

ELIGIBILITY:
Inclusion criteria

1. Women aged 18-40 years
2. Bilateral patent tubes demonstrated by hysterosalpingogram, hysterosalpingo-contrast sonography or laparoscopy
3. Regular menses 21 to 35 days Normal semen parameters :Total motile sperm count ≥10 million. (World Health Organization criteria, 2010)

Exclusion criteria

1. Unwillingness to accept either of the two interventions
2. Contra-indications to acupuncture: pacemaker use or bleeding disorder
3. Received acupuncture before 2 months for other diseases which are not related to unexplained infertility.
4. Previously received acupuncture for unexplained infertility
5. Use of hormonal or other medication (including Chinese Herbal prescriptions) which may affect the outcome in the past 2 months.
6. Patients who anticipate taking longer than a one month break from treatment during the trial (i.e. 4 months from randomization).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1423 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
live birth rate | Up to 4 months

SECONDARY OUTCOMES:
pregnancy rate | Up to 14 months
Miscarriage rate | Up to 14 months
Other pregnancy complications such as early pregnancy loss, gestational diabetes mellitus, pregnancy-induced hypertension and birth of small-for-gestational-age (SGA) babies. | Up to 14 months
quality of life | Up to 14 months
Side effect | Up to 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoke Wu, MD.PhD., Study Chair — The First Affliated Hospital,Heilongjiang University of Chinese Medicine
Locations (16):
- China (16):
  - Guangzhou Medical School First Affiliated Hospital, Guangzhou, Guangdong
  - The Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Daqing Longnan hospital, Daqing, Heilongjiang
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Department of Obstetrics and Gynecology,First Affliated Hospital,Heilongjiang University of Chinese Medicine ., Harbin, Heilongjiang
  - Obstetrics and Gynecology,Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - First Affiliated Hospital of Hunan University of Chinese, Changsha, Hunan
  - Maternal and Child Health Hospital of Xuzhou, Xuzhou, Jiangsu
  - Jiangxi University of Chinese Medicine Affiliated Hospital, Nanchang, Jiangxi
  - First Hospital, Jiangxi college of Chinese Medicine, Nanchang, Jiangxi
  - Shanxi Chinese Medicine Hospital, Shangxi, Shanxi
  - Shanxi Hospital of Chinese Medicine, Taiyuan, Shanxi
  - Tianjin Tanggu Maternity and Child Care Center, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Tianjin University of Chinese Medicine, Tianjin, Tianjin Municipality
  - Wenzhou Chinese Medicine Hospital, Wenzhou, Zhejiang
  - Hangzhou Chinese Medicine Hospital, Hangzhou